CLINICAL TRIAL: NCT03408275
Title: Dietary Patterns and Variability in Blood Lead Concentrations Among Pregnant British Women
Brief Title: Dietry Pattern and Lead Levels in Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Bristol (Other)
Collaborators: Wellcome Trust (Other); Medical Research Council (Other Government); Bristol Biomedical Research Unit (Unknown)
Responsible Party: Sponsor
Other Study IDs: ALSPAC_2
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Dietary Habits; Lead Poisoning; Pregnancy Related
Keywords: Dietary patterns; Pregnancy; Woman; Diet; Lead; ALSPAC
MeSH Terms: conditions — Feeding Behavior; Lead Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women enrolled in ALSPAC
  Interventions: Other: None - observational

INTERVENTIONS:
Other: None - observational — None - observational

SUMMARY:
During pregnancy lead crosses the placenta freely and can have adverse effects on the fetus, with the potential for life-long impact on the child. Identification of dietary patterns and food groups in pregnancy in relation to measures of lead status could provide a more useful alternative to a nutrient-specific advice to minimise fetal exposure to lead during pregnancy. The aim is to evaluate whether dietary patterns and food groups are associated with blood lead concentrations in pregnancy.

DETAILED DESCRIPTION:
Whole blood samples were collected from pregnant women enrolled in the Avon Longitudinal Study of Parents and Children observational birth cohort study and were analysed for lead. Dietary pattern scores were derived from principal components analysis of a food frequency questionnaire. Associations of quartiles of dietary pattern scores, and of food groups categorised by frequency of consumption, with the likelihood of blood lead concentration (B-Pb) ≥5 µg/dl will be identified with adjusted logistic regression (n=2167).

ELIGIBILITY:
Inclusion Criteria: Enrolled in ALSPAC, pregnant -

Exclusion Criteria: Not enrolled in ALSPAC, not pregnant

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The sample for this analysis was derived from the Avon Longitudinal Study of Parents and Children (ALSPAC), which is a UK-based birth cohort set up to investigate environmental and genetic influences on health and disease. ALSPAC recruited 14,541 pregnant women resident in Avon, UK with expected dates of delivery between 1st April 1991 and 31st December 1992.
Sampling Method: Non-Probability Sample
Enrollment: 2167 (Actual)
Dates: Start 1991-04-01 (Actual); Primary Completion 1992-12-01 (Actual); Study Completion 1992-12-01 (Actual)

PRIMARY OUTCOMES:
Blood lead concentration | During gestation
  Blood lead concentration

CONTACTS AND LOCATIONS:
Overall Officials: Nic Timpson, PhD, Study Director — University of Bristol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Individual Participant Data Set — http://www.bristol.ac.uk/alspac/ — ALSPAC data available to researchers on application through the website